CLINICAL TRIAL: NCT03935789
Title: Feasibility of Better Living After Stroke Through Technology
Acronym: BLAST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: University shutdown due to COVID
Sponsor: University of Missouri-Columbia (Other)
Collaborators: BrightOutcome (Industry); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Timothy J Wolf, Associate Professor, Occupational Therapy, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013982; R44NR016183 (NIH)
Record Dates: First submitted 2019-04-25; First posted 2019-05-02 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Stroke
Keywords: stroke; occupational therapy; participation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single group feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BLAST (Experimental): All participants in this study will be assigned to this group to participate in the BLAST intervention. The intervention will be a self-guided web-based platform using a self-management model to help support better engagement in everyday life activity
  Interventions: Behavioral: BLAST

INTERVENTIONS:
Behavioral: BLAST — 12-week self-guided intervention using a web-based platform

SUMMARY:
The investigators propose to evaluate the feasibility of Better Living After Stroke through Technology (BLAST) to help stroke survivors and family members return back to their productive and meaningful lives by proactively 1) helping them set their activity goals using ACS, 2) assessing their behavioral/functional capabilities using FBP, 3) recognizing symptoms indicative potential secondary stroke risks, 4) engaging support from online/community resources, and 5) offering tailored self-management recommendations using evidence-based strategies on how to achieve their activity goals and avoid secondary stroke based on their capabilities, stroke-related symptoms and available social resources.

DETAILED DESCRIPTION:
Stroke, which is the leading cause of disability, cognitive impairment and death in the US, imposes significant financial and personal burden. Although the residual effects of stroke affect many aspects of life, many aspects are not addressed by traditional rehabilitation treatments. In particular, persons with mild stroke, typically defined as a stroke with no or slight motor impairment and a high level of independence in basic activities of daily living, often experience emotional problems, subtle but significant cognitive impairment and decreased participation in productive, social and leisure activity. Despite these problems, persons with mild stroke are typically discharged to home without further referral to health or rehabilitation services other than follow-up with primary care physicians.

This application is in response to RFA PA-11-335 (Lab to Marketplace: Tools for Biomedical and Behavioral Research), a special 2-year Phase I SBIR program to accelerate the translation of behavioral research from academic to the marketplace. The project is based on the extensive research that developed and tested reliable and valid measures of activity participation (Activity Card Sort, or ACS) and cognitive skills supporting performance of simple and complex functional tasks (Functional Behavior Profile, or FBP). These measures have been used to guide treatments to help persons with mild cognitive impairment and their families support functional independence. These measures and the results of other studies will be used to build a dynamic online self-management tool designed to help persons with mild stroke develop individualized strategies that will support optimal recovery.

The investigators propose to evaluate the feasibility of Better Living After Stroke through Technology (BLAST) to help stroke survivors and family members return back to their productive and meaningful lives by proactively 1) helping them set their activity goals using ACS, 2) assessing their behavioral/functional capabilities using FBP, 3) recognizing symptoms indicative potential secondary stroke risks, 4) engaging support from online/community resources, and 5) offering tailored self-management recommendations using evidence-based strategies on how to achieve their activity goals and avoid secondary stroke based on their capabilities, stroke-related symptoms and available social resources.

Stroke survivors and family using the BLAST system are expected to have 1) better life satisfaction as measured by the Overall Recovery item of the Stroke Impact Scale; 2) increased activity as measured by Activity Card Sort; 3) better problem-solving and task performance as measured by Functional Behavior Profile; and 4) fewer caregiver concerns as measured by the Stroke Caregiver Needs Scale.

Specific Aims: 1) to evaluate the acceptability of BLAST ; and 2) to evaluate the preliminary effect of BLAST on self-efficacy, participation, and community reintegration.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age and older
* diagnosis of mild to moderate ischemic stroke (NIHSS <16)
* 3 months to 5 years post-stroke onset (of most recent stroke)
* the availability of a willing caregiver or supportive individual throughout the intervention
* access to a computer or tablet with internet access
* discharged from the hospital to the community
* able to read, write, and speak English fluently; and (8) community dwelling

Exclusion Criteria:

* history of functional impairment prior to the index stroke as self-reported on the Telephone Screening Form
* current diagnosis of a severe psychiatric disorder
* current drug/alcohol abuse
* terminal illness
* Montreal Cognitive Assessment score of less than 23
* direct verbal cue required for EFPTe test
* severe depressive symptoms as indicated on the Patient Health Questionnaire (PHQ-9 score greater than 19)
* any thoughts of harming themselves or others as indicated on question #9 of the PHQ-9.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
Participation Strategies Self-Efficacy Scale (change) | Change from baseline score at 12 weeks (post-intervention)
  35-item scale designed to assess self-efficacy in using participation strategies following a stroke using six subscales: (1) managing home participation, (2) staying organized, (3) planning and managing community participation, (4) managing work/productivity, (5) managing communication, and (6) advocating for resources, where higher scores equate to more self-efficacy.
Activity Card Sort (change) | Change from baseline score at 12 weeks (post-intervention)
  records the activity participation and engagement of adults in instrumental, leisure and social activities currently and prior to a health event. Possible scores 0 - 32 where 32 indicates the most activity.
Patient-Reported Outcomes Measurement Information System (PROMIS)- 29 (change) | Change from baseline score at 12 weeks (post-intervention)
  generic health-related quality of life survey, assesses each of the 7 PROMIS domains: depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; and ability to participate in social roles and activities. Scale of 1 - 5, where 1 = poorest quality of life and 5 = best quality of life.
Stroke Impact Scale (change) | Change from baseline score at 12 weeks (post-intervention)
  stroke-specific, self-report, health status measure. It was designed to assess multidimensional stroke outcomes, including strength, hand function Activities of Daily Living / Instrumental Activities of Daily Living, mobility, communication, emotion, memory and thinking, and participation. Total possible score = 59 - 295 where 295 = the least impact of stroke.
After Scenario Questionnaire | 12-weeks after baseline assessment (post-intervention)
  assessment of acceptability of the intervention. Scale of 1 - 7 where 1 = lowest acceptability and 7 = most acceptability.
Post Study System Usability Questionnaire | 12-weeks after baseline assessment (post-intervention)
  assessment of participant satisfaction and evaluation of usability of the web-based platform. Scale of 1 - 7 where 1 = least satisfaction and 7 = most satisfaction.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) (change) | Change from baseline score at 12 weeks (post-intervention)
  9-item depression scale. Total possible score = 0 - 27 where 0 = no depression and 27 = severe depression.
Executive Function Performance Test- Enhanced (EFPTe) (change) | Change from baseline score at 12 weeks (post-intervention)
  assessment tool used to measure executive functioning in daily life activities. Scale of 0 - 5 where 0 = most independence and 5 = least independence.
Functional Behavior Profile (change) | Change from baseline score at 12 weeks (post-intervention)
  clinical assessment measure that provides caregivers with a method of describing the impaired person's capabilities in performing tasks, social interactions, and problem-solving following a stroke. Total possible score = 0 - 108 where 108 = most functional behavior.
Reintegration to Normal Living Index/Scale (change) | Change from baseline score at 12 weeks (post-intervention)
  assessment of the degree to which individuals who have experienced traumatic or incapacitating illness achieve reintegration into normal social activities (e.g. recreation, movement in the community, and interaction in family or other relationships). Total possible score = 0 - 100 where 100 = total reintegration.
Lawton Instrumental Activities of Daily Life Scale (change) | Change from baseline score at 12 weeks (post-intervention)
  assessment for identifying how a person is functioning at the present time and for identifying improvement or deterioration over time in IADL activities. Total possible score = 0 - 8 where 8 = high function.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Wolf, OTD, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri: Department of Occupational Therapy, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No